CLINICAL TRIAL: NCT03977883
Title: Management of Paroxystic Atrial Fibrillation in French Intensive Care Units
Acronym: PAF-ICU
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: French Society of Anesthesia and Intensive Care Medecine (Unknown)
Responsible Party: Sponsor
Other Study IDs: PAF-ICU - RNI 2018 CONSTANTIN
Record Dates: First submitted 2019-05-29; First posted 2019-06-06 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: New Onset Atrial Fibrillation; ICU Patients
Keywords: New onset atrial fibrillation; Paroxystic atrial fibrillation; ICU patients; Rate control; Rhythm control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose of the study is to evaluate treatment of new onset atrial fibrillation in french ICU.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common arrhythmia in the ICU and is associated with significant morbidity. However, curative treatment remains unclearly established. In fact, there are no specific recommendations for new onset atrial fibrillation in ICU and only few studies have assessed this topic.

The PAF-ICU trial is an observational, prospective, multicenter, transversal trial. The main objective is to evaluate the management of paroxytic atrial fibrillation that occur in ICU.

The investigators want to document 2500 episodes of paroxystic atrial fibrillation in 50 ICU centers. In each center, the episodes are included consecutively until the required 50 episodes are obtained for each center.

A patient can present several episodes and each episode can be included in the study. A new episode is considered as such if it occurs more than one hour after the previous episode.

The follow-up period for each patient corresponds to the ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient hospitalized in ICU
* New onset atrial fibrillation

Exclusion Criteria:

* Age < 18 years
* Parturient or breast-feeding woman
* Persistent or permanent atrial fibrillation
* Patients after cardiovascular or thoracic surgery
* Patients with therapeutic limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in French ICU
Sampling Method: Non-Probability Sample
Enrollment: 742 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Management of Atrial Fibrillation | ICU stay (until 28 days)
  All types of therapeutics used to manage atrial fibrillation are collected

SECONDARY OUTCOMES:
Cardiac rhythm status | Before, 5 minutes, 30 minutes, 1 hour, and 24 hours after atrial fibrillation
  Type of rhythm : Normal (sinus rhythm), Atrial Fibrillation, Other disturbance
Blood pressure | Before, 5 minutes, 30 minutes, 1 hour, and 24 hours after atrial fibrillation
  Blood pressure. Unit : Millimeters of mercury
Heart rate | Before, 5 minutes, 30 minutes, 1 hour, and 24 hours after atrial fibrillation
  Heart rate. Unit : beats per minute
Cardiac output | Before, 5 minutes, 30 minutes, 1 hour, and 24 hours after atrial fibrillation
  Product of the heart rate (HR) and the stroke volume (SV), which is the volume of blood pumped from the ventricle per beat. Unit : L/min.
ScvO2 | Before, 5 minutes, 30 minutes, 1 hour, and 24 hours after atrial fibrillation
  Venous saturation. Unit : percentage
Vasopressors | Before, 5 minutes, 30 minutes, 1 hour, and 24 hours after atrial fibrillation
  Type of vasopressors used
Stroke | ICU Stay up to 28 days
  Occurrence of stroke during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Constantin, Study Director — Réa Adulte CHU Clermont-Ferrand; Bernard Cosserant, Principal Investigator — Neuro-Réa CHU Clermont-Ferrand; Raiko Blondonnet, Principal Investigator — RMC CHU Clermont-Ferrand; Eric Kipnis, Principal Investigator — CHU Lille; Jonathan Paillot, Principal Investigator — CHU Besancçon; Charles Vidal, Principal Investigator — CHU de la Réunion; Laurent Muller, Principal Investigator — CHU Nimes; Johann Auchabie, Principal Investigator — CH Cholet; Guillaume Grillet, Principal Investigator — CH Lorient; Philippe Seguin, Principal Investigator — CHU Rennes; Philippe Guerci, Principal Investigator — CHRU Nancy; Bernard Lalanne, Principal Investigator — Hôpital Saint-Joseph - Marseille; Marc Leone, Principal Investigator — Hôpital Nord - APHM; Stanislas Ledochowski, Principal Investigator — CH Bourgoin-Jallieu; Matthieu Legrand, Principal Investigator — Hôpital Saint-Louis - APHP; Jeremy Bourenne, Principal Investigator — La Timone APHM; Michel Durand, Principal Investigator — University Hospital, Grenoble; Antoine Monsel, Principal Investigator — La Pitié Sapêtrière; Mathieu Guilbart, Principal Investigator — CHU Amiens; Matthieu Biais, Principal Investigator — University Hospital, Bordeaux; Cédric Bruel, Principal Investigator — CH Saint-Joseph Paris; Antoine Roquilly, Principal Investigator — Nantes University Hospital; Gaëtan Plantefeve, Principal Investigator — CH Argenteuil; Jérôme Morel, Principal Investigator — CHU SAINT-ETIENNE; Carole Ichai, Principal Investigator — CHU NICE; Adrien Auvet, Principal Investigator — CH Dax; Enora Atchade, Principal Investigator — Hôpital Bichat; Sigismond Lasocki, Principal Investigator — University Hospital, Angers; Pierre-Eric Danin, Principal Investigator — Clinique Les Sources Nice; Marc Danguy Des Deserts, Principal Investigator — Hôpital d'Instruction des Armées de Brest; Evelina Ochin Salatova, Principal Investigator — Hôpital Simone Veil - CH d'Eaubonne; Antoine Rouget, Principal Investigator — University Hospital, Toulouse; Armand Mekontso Dessap, Principal Investigator — Hôpital Henri Mondor APHP; Justine Perrot, Principal Investigator — CHU Dijon; Jibba Amraoui, Principal Investigator — Institut Régional du Cancer de Montpellier; Matthias Garot, Principal Investigator — CHU Lille
Locations (32):
- France (32):
  - CHU, Amiens
  - CHU, Angers
  - CH, Argenteuil
  - CHU, Besançon
  - CHU, Bordeau
  - CH, Bourgoin
  - Hôpital d'Instruction des Armées, Brest
  - CH, Cholet
  - CHU, Clermont-Ferrand
  - CH, Dax
  - CHU, Dijon
  - CH, Eaubonne
  - CHU, Grenoble
  - CHU, Lille
  - Hôpital du Scorff, Lorient
  - APHM, Marseille
  - Hôpital Saint-Joseph, Marseille
  - La Timone APHM, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - CHU, Nancy
  - CHU, Nantes
  - CHU, Nice
  - Clinique médicale les Sources, Nice
  - CHU, Nîmes
  - Groupe Hospitalier Saint Joseph, Paris
  - Hôpital Bichat, Paris
  - Hôpital Henri Mondor, Paris
  - Hôpital La Pitié Salpêtrière, Paris
  - Hôpital Saint-Louis, Paris
  - CHU, Rennes
  - CHU, Saint-Etienne
  - CHU, Toulouse

REFERENCES:
- [Derived] Pardo E, Futier E, Muller L, Besch G, Vardon-Bounes F, Kipnis E, Lasocki S, Ledochowski S, Ochin E, Bourenne J, Grillet G, Auvet A, Mekontso Dessap A, Bruel C, Launey Y, Fiorillo M, Jabaudon M, Godet T, Mulliez A, Constantin JM; SFAR Research Network. Management of new-onset atrial fibrillation in critically ill patients: A national multicenter prospective cohort. Anaesth Crit Care Pain Med. 2026 Jan;45(1):101617. doi: 10.1016/j.accpm.2025.101617. Epub 2025 Sep 26. PMID 41016469